CLINICAL TRIAL: NCT03578198
Title: Phase II Study of Rituximab Plus MG4101 in Patients With Relapsed or Refractory Indolent CD20-positive Non-Hodgkin Lymphoma (NHL)
Brief Title: Rituximab Plus MG4101 Indolent CD20-positive Non-Hodgkin Lymphoma (NHL)
Acronym: MG4101
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Issues in supply of IP
Sponsor: Seoul National University Hospital (Other)
Collaborators: Hallym University Medical Center (Other); Kyunghee University Medical Center (Other); Gyeongsang National University Hospital (Other)
Responsible Party: Principal Investigator, Tae Min Kim, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Truximab+MG4101
Record Dates: First submitted 2018-06-25; First posted 2018-07-06 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: CD20-positive Non-Hodgkin Lymphoma
MeSH Terms: interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rituximab + MG4101 (Experimental): Drug: Rituximab + MG4101
  Induction phase:
  Rituximab (Truxima) 375mg/m2 IV Weekly (X4) MG4101 3x107 cells/kg IV Weekly (X4) Maintenance phase
  Rituximab (Truxima) 375mg/m2 IV q 4 weeks (X4) MG4101 3x107 cells/kg IV q 4 weeks (X4)
  Interventions: Drug: Rituximab + MG4101

INTERVENTIONS:
Drug: Rituximab + MG4101 — 1. Induction phase:
     * Rituximab (Truxima) 375mg/m2 IV Weekly (X4)
     * MG4101 3x107 cells/kg IV Weekly (X4)
  2. Maintenance phase
     * Rituximab (Truxima) 375mg/m2 IV q 4 weeks (X4)
     * MG4101 3x107 cells/kg IV q 4 weeks (X4)

SUMMARY:
Phase II study of rituximab plus MG4101 in patients with relapsed or refractory indolent CD20-positive non-Hodgkin lymphoma (NHL) Investigator-Initiated Trials

DETAILED DESCRIPTION:
Multi-center trial, Phase II, non-randomized, open-label, single-arm study with combined therapy of rituximab plus MG4101 in patients with indolent CD20-positive NHLs who has relapsed or refractory to prior chemotherapy or chemo-radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed indolent CD20-positive NHLs (iNHLs; follicular lymphoma grade 1-3a, marginal zone B-cell lymphoma, small lymphocytic lymphoma, Waldenstrom macroglobulinemia)
2. CD20-positive iNHL patients who relapsed or progressed
3. ≥ 19 years
4. ECOG PS 0-2
5. At least one bidimensionally measurable disease (or presence of IgM paraproteinemia ≥ 2 x ULN for Waldenstrom macroglobulinemia)
6. Adequate hematologic, renal, and hepatic functions
7. Appropriate methods of contraception during the study
8. Written informed consent

Exclusion Criteria:

1. Not all of the above inclusion criteria are met.
2. Prior chemotherapy within 4 weeks or radiotherapy within 6 weeks
3. Corticosteroids > 10mg/day during last 28 days
4. Evidence of CNS involvement by lymphomas
5. Active HBV/HCV infections, known HIV infection
6. Prior diagnosis of cancers within 5 years
7. Serious concurrent cardiovascular disease
8. Patients who are pregnant or lactating

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-11-08 (Actual); Primary Completion 2022-04-07 (Actual); Study Completion 2022-04-07 (Actual)

PRIMARY OUTCOMES:
Overall response rate | Through treatment completion, an average of 25 weeks
  Investigator-assessed, confirmed objective response by revised response criteria

SECONDARY OUTCOMES:
Complete remission rate | Through treatment completion, an average of 25 weeks
  Confirmed complete remission by revised response criteria
Progression-free survival | From date of initiation until the date of first documented progression, whichever came first, assessed up to 2 years
  PFS as defined by revised response criteria
Overall survival | Through study completion, an average of 2 years
  OS as defined by revised response criteria

CONTACTS AND LOCATIONS:
Overall Officials: Tae Min Kim, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No